CLINICAL TRIAL: NCT06261034
Title: Sex Differences in Neurocirculatory Control With Obstructive Sleep Apnea
Brief Title: A Study of Sex Differences in Neurocirculatory Control
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Joshua M. Bock, Principal Investigator, Mayo Clinic
Other Study IDs: 23-008765; 8K12AR084222-15 (NIH)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to investigate potential sex differences in neurocirculatory control of blood pressure in patients with untreated obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years of age

Exclusion Criteria:

* Coronary artery disease
* Heart failure
* Pregnancy
* COPD
* Diabetes
* CKD
* Sleep disorders other than OSA
* Shift workers
* Individuals who typically go to sleep after midnight
* Individuals who traveled across ≥2 time zones within one week of study visits
* BMI ≥40.0kg/m2
* Use of nicotine-containing products within the two years preceding study visits
* Use of allopurinol, proton pump inhibitors, or other medications/supplements which interfere with outcome measures

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with or without untreated obstructive sleep apnea will be recruited from Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Baseline
  Measured in millimeters of mercury (mmHg).
Arterial stiffness | Baseline
  Measured by applanation tonometry reported as aortic pulse wave velocity (m/sec)
Endothelial function | Baseline
  Ultrasound assessment of flow-mediated vasodilation of the brachial artery. Brachial artery diameter and blood velocity will be measured after deflation to measure endothelial function.

SECONDARY OUTCOMES:
Sympathetic nerve burst frequency | Baseline
  Measured by Microneurography reported as number of nerve bursts per minute (burst/min)
Sympathetic nerve burst incidence | Baseline
  Measured by Microneurography reported as number of nerve burst per 100 heart beats (burst/100 heart beats)
Sympathetic nerve burst amplitude (AU) | Baseline
  Measured by Microneurography reported in arbitrary units (AU)
Total muscle sympathetic nerve activity (MSNA) | Baseline
  Measured by Microneurography reported burst arbitrary units per minute (AU/min)

OTHER OUTCOMES:
Cerebral autoregulation | Baseline
  Measured by transcranial doppler ultrasound (cm/sec).
Sympathetic action potentials per burst | Baseline
  Measured by Microneurography reported as action potentials per burst (reflecting firing rate).
Sympathetic action potential clusters per burst | Baseline
  Measured by Microneurography reported as clusters per burst (reflecting recruitment of latent subpopulations).
Sympathetic action potential conduction latency of each cluster | Baseline
  Measured by Microneurography reported as conduction latency of each cluster (reflecting synaptic delays and verifying larger amplitude clusters as new populations).
Immune function | Baseline
  Immune function will be measured as percent of parent cell population.
Urinary Extracellular Vesicle Presence and Content | Baseline
  Number of extracellular vesicles present in a 24 hour urine collection and the contents being carried by those vesicles.
Plasma Extracellular Vesicle Presence and Content | Baseline
  Number of extracellular vesicles present in blood plasma sample and the contents being carried by those vesicles.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Bock, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No